CLINICAL TRIAL: NCT07272109
Title: Active Anti-diabetic Treatment Plus Chemotherapy for Metastatic Pancreatic Cancer Related Diabetes Mellitus (Type 3c)
Brief Title: Active Anti-diabetic Treatment Plus Chemotherapy for Pancreatic Cancer Related Diabetes
Acronym: PTCA199-16
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Guopei Luo, Prof., Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTCA199-16
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer
Keywords: diabetes melltus; metastatic pancreatic cancer; type 3c
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Hypoglycemic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active anti-diabetic treatment (Experimental)
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine (1000 mg/m2); Other: Anti-Diabetics; Other: Active treatment and monitoring
- Regular anti-diabetic treatment (Active Comparator)
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine (1000 mg/m2); Other: Anti-Diabetics

INTERVENTIONS:
Drug: Nab-paclitaxel — 120 mg per square meter of body-surface area on days 1, 8, and 15 every 4 weeks
Drug: Gemcitabine (1000 mg/m2) — (1000 mg per square meter) on days 1, 8, and 15 every 4 weeks
Other: Anti-Diabetics — Metformin, insulin or other anti-diabetic treatments
Other: Active treatment and monitoring — Attend follow-ups at designated endocrinology clinics, with proactive inquiry about hypoglycemic measures and medication implementation.
  Arms: Active anti-diabetic treatment

SUMMARY:
The purpose of this study is to evaluate the efficacy of anti-diabetic treatment on improving the overall survival for metastatic pancreatic cancer patients complicated by diabetes receiving gemcitabine and nab-paclitaxel chemotherapy.

DETAILED DESCRIPTION:
About 80% of patients with pancreatic adenocarcinoma have aberrant fasting blood glucose at the time of diagnosis. The consistent association between pancreatic cancer and diabetes mellitus has long been recognized and even been termed as "chicken and egg". Many reports have found that pancreatic cancer can result in diabetes, which is called type 3c diabetes. New-onset diabetes is commonly observed in pancreatic cancer patients and has been considered as a potential screening sign. Moreover, diabetes has been found as a predictor of poor outcome in pancreatic cancer.

Pancreatic cancer cells have a strong dependence on glucose and they are well-known for their sweet teeth. High glucose is associated with impaired immunologic reaction, intolerability to chemotherapy, radiotherapy and other major treatments, an increased risk of pancreatic surgery. Given the linkage between pancreatic cancer and diabetes or high blood glucose, a clinical trial is needed to validate the effect of anti-diabetic treatment in type 3c diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Age ≥ 18 years and ≤ 80 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Histologically or cytologically confirmed metastatic pancreas adenocarcinoma.
* History of diabetes mellitus, or newly diagnosed diabetes meeting the diagnostic criteria of the American Diabetes Association.
* The expected survival ≥ 3 months.
* Able to comply with study visit schedules and other protocol requirements.

Exclusion Criteria:

* • History of other malignancies requiring anti-cancer therapy within 2 years prior to enrollment (except treated Stage I prostate cancer, in situ cervical cancer, in situ breast cancer, etc.);

  * Non-primary pancreatic cancer patients;
  * Digestive tract inflammation, including biliary tract infection, gastrointestinal infection, pancreatitis, etc.;
  * Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS): | 2 months
  Time from randomization to death from any cause

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 months
  Time from enrollment to first tumor progression.
Blood Glucose Control | One month
  Changes in fasting blood glucose levels.
Rate of HbA1c Control | One month
  Changes in glycated hemoglobin compared to baseline.

OTHER OUTCOMES:
Serum Tumor Marker Changes: | One month
  Changes in CA19-9, CEA, and CA125 levels compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Guopei Luo, MD, Study Chair — Shanghai Cancer Center
Locations (1):
- Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhu X, Xiao Z, Liu H, Zhang P, Deng S, Ding L, Feng J, Luo J, Ni Q, Luo G, Yu X. Pancreatic Cancer: An Exocrine Tumor With Endocrine Characteristics. Ann Surg. 2024 Dec 1;280(6):e17-e25. doi: 10.1097/SLA.0000000000006168. Epub 2023 Dec 5. PMID 38050737